CLINICAL TRIAL: NCT03925155
Title: A Randomized Trial to Investigate if a Pre-operative Wash With Chlorhexidine vs Povidone-iodine Vaginal Scrub Decreases Infectious Morbidity in Patients Undergoing Cesarean Section After Ruptured Membranes
Brief Title: RCT Investigating Pre-cesarean Vaginal Wash of Chlorhexidine vs Povidone-iodine for Patient With Ruptured Amniotic Membrane.
Acronym: VAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn from the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Meleen Chuang, Assistant Professor, MD FACOG, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-9948
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Cesarean Section Complications
Keywords: vaginal prep; randomization; chlorhexidine; povidone iodine
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Intervention Model Description: One arm is standard of care 10% povidone-iodine preparation, comparing with trial of chlorhexidine 4% vaginal preparation
Who Masked: Participant
Masking Description: Participants will be blinded to the arm in which they have been assigned. Providers will need to perform vaginal preparation and solutions look different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chlorhexidine gluconate vaginal scrub (Experimental): Use of chlorhexidine 4% vaginal scrub instead of current standard of care 10% povidone iodine vaginal scrub for cesarean sections
  Interventions: Drug: EZ scrub vaginal chlorhexidine 4% solution
- Povidone-iodine vaginal scrub (Active Comparator): Current standard of care 10% povidone iodine vaginal scrub for cesarean sections
  Interventions: Drug: 10% provodine-iodine vaginal preparation

INTERVENTIONS:
Drug: EZ scrub vaginal chlorhexidine 4% solution — Patients will be randomized to receive one of two solutions. Either chlorhexidine 4% solution or standard of care 10% provodine-iodine vaginal solution
  Other Names: vaginal preparation using providone iodine
  Arms: Chlorhexidine gluconate vaginal scrub
Drug: 10% provodine-iodine vaginal preparation — Patients will be randomized to receive one of two solutions. Either chlorhexidine 4% solution or standard of care 10% provodine-iodine vaginal solution
  Arms: Povidone-iodine vaginal scrub

SUMMARY:
The objective of this study is to investigate if the rate of infectious morbidity is decreased with the use of chlorhexidine or povidone-iodine vaginal scrub before cesarean section after ruptured membranes.

DETAILED DESCRIPTION:
Postpartum endometritis is an infection of the endometrial lining of the uterus clinically diagnosed by fever and uterine fundal tenderness. The most important risk factor for developing endometritis is cesarean section, as it occurs in 11% of cesarean sections after labor and 3% of elective cesarean sections. Other risk factors for endometritis are chorioamnionitis, prolonged labor, prolonged rupture of membranes and vaginal colonization with Group B Streptococcus. Some complications of endometritis include prolonged hospital stay, sepsis, peritonitis and intrapelvic abscess.

Surgical site infections are infections of the incision, organ or space after a procedure and are responsible for 38% of infections in patients undergoing surgery. In obstetric patients, infectious morbidity (wound complication, surgical site infections, endometritis) occurs in 5-10% of cesarean sections, which is 5-fold higher than vaginal deliveries. Additionally, infectious morbidity is thought to be highest in those patients who have cesarean sections after undergoing labor.

Current practices endorsed by ACOG and the CDC to reduce the incidence of infectious morbidity after cesarean section include pre-operative antibiotics and pre-operative skin cleansing with chlorhexidine skin preparation. Chlorhexidine and povidone-iodine are chemical antiseptics that reduces bacteria found on the skin. Additionally, vaginal scrub with 4% chlorhexidine gluconate and 10% povidone-iodine antiseptic solution immediately prior to cesarean section has been embraced into some practices as a means to decrease infectious morbidity. There is abundant literature showing pre-operative vaginal cleansing prior to hysterectomy has been shown to decrease vaginal surgical site antisepsis, however research on its use prior to cesarean section is limited.

This study aims to assess the effectiveness of pre-operative vaginal scrub with 4% chlorhexidine or 10% povidone iodine in reducing infectious morbidity (specifically endometritis and SSI) in patients undergoing cesarean section with previously ruptured membranes. Current standard of care is use of pre-operative vaginal scrub with 10% povidone iodine. Patients will be randomized to one of two groups using pre-operative vaginal scrub for 30 seconds: 4% chlorhexidine or 10% povidone iodine. In addition both groups will receive pre-operative antibiotics with cefazolin and azithromycin, as well as abdominal cleansing with chlorhexidine-alcohol based skin preparation and 0.25% chlorhexidine wipe for 30 seconds, as this is standard of care for women undergoing cesarean section with ruptured membranes. In the event of penicillin allergy, antibiotics are adjusted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-50 years
* The study will be offered to women at > 24 weeks gestation who are undergoing nonemergent cesarean delivery with ruptured amniotic membranes.
* All patients undergoing cesarean delivery with ruptured amniotic membranes.

Exclusion Criteria:

* Minors
* Emergent cesarean delivery.
* No ruptured membranes.
* Allergy to chlorhexidine or povidone-iodine.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Endometritis | 30 day postoperative
  determine if there is any change of rates of postpartum endometritis amongst the chlorhexidine vaginal preparation group compared to povidone iodine group

SECONDARY OUTCOMES:
Rate of wound complications | 30 day postoperative
  Change of wound complication among postpartum 30 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Meleen Chuang, MD, Study Chair — Montefiore Medical Center, Dept OB/GYN

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed MR, Aref NK, Sayed Ahmed WA, Arain FR. Chlorhexidine vaginal wipes prior to elective cesarean section: does it reduce infectious morbidity? A randomized trial. J Matern Fetal Neonatal Med. 2017 Jun;30(12):1484-1487. doi: 10.1080/14767058.2016.1219996. Epub 2016 Sep 1. PMID 27583685
- [Result] Haas DM, Morgan S, Contreras K, Enders S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2018 Jul 17;7(7):CD007892. doi: 10.1002/14651858.CD007892.pub6. PMID 30016540
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895